CLINICAL TRIAL: NCT03077230
Title: Pre-Post Study for Supporting Appropriate Implementation of Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC 1506
Record Dates: First submitted 2016-11-22; First posted 2017-03-10 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Lung Neoplasms; Early Detection of Cancer; Decision Support Techniques; Primary Health Care
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre/Post Test of a Lung Cancer Screening Decision Aid (Experimental)
  Interventions: Behavioral: Pre/Post Test of a Lung Cancer Screening Decision Aid

INTERVENTIONS:
Behavioral: Pre/Post Test of a Lung Cancer Screening Decision Aid — After completing the baseline survey, the research team member will ask each participant asked to view the lung cancer screening decision aid on a tablet. The following areas regarding lung cancer screening: What is lung cancer?, Why is lung cancer a problem?, What is screening?, What is low-dose CT screening, Recommended frequency of screening, Screening factors, lung cancer risks and benefits (magnitude of benefit, harms, false positive, invasive procedures, radiation, stress/anxiety), Summary, Values Clarification, Screening Choice, and Smoking cessation messaging for current smokers OR positive reinforcement for former smokers.

SUMMARY:
The primary objective of this study is to assess the effect of the decision aid on measures of decision-making such as knowledge, screening attitudes, decisional conflict, and screening intent.

DETAILED DESCRIPTION:
Using a single group, pre-post design, we aim to assess the effect of the decision aid on screening knowledge, screening attitudes, decisional conflict, and screening intent within 3 months of decision aid viewing.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in this study:

* Age 55 - 80;
* Current smoker, or former smoker who has less than a 16-year quit history;
* Have at least a 30-pack year smoking history (average packs per day * years smoking); and
* Patient of the Internal Medicine Clinic at University of North Carolina Health Care.

Exclusion Criteria:

All subjects meeting any of the following exclusion criteria at baseline will be excluded from study participation:

* Ever diagnosed with lung cancer;
* Undergone chemotherapy or radiation therapy in the past 18 months prior to enrollment;
* Coughed up blood from lungs (also called hemoptysis) within the past year prior to enrollment;
* Experienced unexplained weight loss of 15-pounds or more during six months prior to enrollment; and
* Had a chest CT scan within the past 18 months prior to enrollment.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in decision-making measures of knowledge | At time of intervention
  We will use descriptive statistics to provide an overview of knowledge at baseline and at follow-up.
  * Hypothesis 1: Screening specific knowledge will improve after completing the decision aid.
    o Statistical tests:
  * Overall knowledge: Treating knowledge as a continuous variable by adding number correct out of 12 items (0-12 possible points), we will perform a Wilcoxon sign rank test to assess change in knowledge between baseline and follow-up
  * Individual knowledge items: Using McNemar's test, we will compare the proportion who correctly answered individual knowledge items at baseline and follow-up
Change in screening attitudes | At time of intervention
  We will use descriptive statistics to provide an overview of screening attitudes at baseline and at follow-up.
  • Exploratory: Using t-tests or chi-squared tests as appropriate, we will assess the change between baseline and follow-up of screening attitudes.
Change in decisional conflict | At time of intervention
  We will use descriptive statistics to provide an overview of decisional conflict at baseline and at follow-up.
  • Exploratory: Using t-tests or chi-squared tests as appropriate, we will assess the change between baseline and follow-up of decisional conflict.
Change in screening intentions | At time of intervention
  We will use descriptive statistics to provide an overview of screening intentions at baseline and at follow-up.
  • Exploratory: Using t-tests or chi-squared tests as appropriate, we will assess the change between baseline and follow-up of screening intentions.

SECONDARY OUTCOMES:
Preliminary estimates on the effect of the decision aid on behavioral outcomes | Within 3 months of intervention
  We will use descriptive statistics (means and proportions) to provide preliminary estimates on the effect of the decision aid on documentation of shared decision-making in the electronic health record and screening behavior at 3 months.
Feasibility of implementing a decision aid intervention in a primary care clinic setting | Through study completion, an average of 1 year
  This is a descriptive and qualitative aim. We will describe measures of feasibility related to time needed to complete surveys, participant ability to navigate decision aid website, number of times assistance is needed to complete surveys/navigate the decision aid website, and type of assistance required.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reuland, MD MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Ambulatory Care Center Internal Medicine Clinic, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Kovalchik SA, Tammemagi M, Berg CD, Caporaso NE, Riley TL, Korch M, Silvestri GA, Chaturvedi AK, Katki HA. Targeting of low-dose CT screening according to the risk of lung-cancer death. N Engl J Med. 2013 Jul 18;369(3):245-254. doi: 10.1056/NEJMoa1301851. PMID 23863051
- [Background] Bach PB, Gould MK. When the average applies to no one: personalized decision making about potential benefits of lung cancer screening. Ann Intern Med. 2012 Oct 16;157(8):571-3. doi: 10.7326/0003-4819-157-8-201210160-00524. No abstract available. PMID 22893040
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for lung cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 4;160(5):330-8. doi: 10.7326/M13-2771. PMID 24378917
- [Derived] Reuland DS, Cubillos L, Brenner AT, Harris RP, Minish B, Pignone MP. A pre-post study testing a lung cancer screening decision aid in primary care. BMC Med Inform Decis Mak. 2018 Jan 12;18(1):5. doi: 10.1186/s12911-018-0582-1. PMID 29325548
- See also: UNC Lineberger Home Page — http://unclineberger.org